CLINICAL TRIAL: NCT02355691
Title: Improvement in Wound Healing With Negative Pressure Wound Therapy for Postoperative Total Hip Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of Personnel
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-1920
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Complications; Arthroplasty, Infection or Inflammation; Wound Complication
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PREVENA Group (Experimental): Patients will be treated with the PREVENA negative pressure device following total hip arthroplasty. This dressing will be used for a period of seven days.
  Interventions: Device: PREVENA
- Standard group (No Intervention): Patients will be treated with the standard absorptive dressing following total hip arthroplasty.

INTERVENTIONS:
Device: PREVENA — The device is a sealed negative pressure wound therapy tool. The device will be placed on the skin during surgery and left in place until their followup at 7 days.
  Other Names: KCI PREVENA Incision Management system
  Arms: PREVENA Group

SUMMARY:
For the target population of adult patients following primary total hip arthroplasty, the randomized clinical trial will be used to evaluate the efficacy of the use of a mobile negative pressure wound therapy(NPWT) device compared to a standard absorptive dressing in the immediate postoperative period. We will apply two dressing types and evaluate the postoperative wounds with a wound scoring system (ASEPSIS) that incorporates multiple variables of wound infection risk.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients undergoing primary total hip arthroplasty.

Exclusion Criteria:

* age less than 18 y/o
* Total hip arthroplasty for fracture
* Revision or conversion total hip arthroplasty
* inability to personally consent to participation due to cognitive impairment, intoxication or sedation
* multiple surgical procedures
* Patients taking immune modulating medication(prednisone, methotrexate, anakinra, etc.)
* skin hypersensitivity to acrylic adhesive or silver.
* Inability to care for dressing due to physical or mental incapacitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Del Gaizo, MD, Principal Investigator — UNC Orthopaedics
Locations (1):
- UNC Orthopaedics, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: PREVENA website — http://www.kci1.com/KCI1/prevena

RESULTS

PARTICIPANT FLOW:
Groups:
- PREVENA Group: Patients will be treated with the PREVENA negative pressure device following total hip arthroplasty. This dressing will be used for a period of seven days.
  PREVENA: The device is a sealed negative pressure wound therapy tool. A single device is placed on the wound at the time of surgery. And removed at the time of the first postop visit around 7 days after surgery.
Period: Overall Study
Arm/Group | PREVENA Group | Standard Group
Started | 7 | 9
1st Postop Visit | 7 | 9
2nd Postop Visit | 7 | 9
Completed | 0 | 0
Not Completed | 7 | 9
Not completed — Loss of Research Personnel | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PREVENA Group | Standard Group | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Full Range); unit: years] | 54.6 [50 to 64] | 57.6 [44 to 73] | 56.2 [44 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 16
Discharge location [Count of Participants; unit: Participants]
  Skilled Nursing Facility | 2 | 3 | 5
  Home | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Wound Healing Scores by the ASEPSIS Criteria
Description: A method of evaluating wounds for infection risk that incorporates multiple wound healing factors such as erythema, drainage, and dehiscence is the ASEPSIS (Additional treatment, presence of Serous discharge, Erythema, Purulent exudate, Separation of the deep tissue, Isolation of bacteria, and duration of inpatient Stay) wound scoring system. Originally developed and validated for cardiac surgery sternal wounds, ASEPSIS evaluates the wound for the severity of multiple factors linked with surgical site infection. This includes dehiscence, exudate/discharge, and erythema. The higher the score, the more likely a surgical site infection will be present. This score will give us a more diverse picture of postoperative wound healing and the influence of Negative Pressure Wound Therapy. Scores can range from 0 to 65, with most scores expected at the lower scale.
Time Frame: (Single point evaluation)-2 weeks post surgery visit
Population: Measured outcomes for all patients that completed the treatment
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | PREVENA Group | Standard Group
Number analyzed (Participants) | 7 | 9
units on a scale | 0.57 [0 to 1] | 1.66 [0 to 16]

2. Secondary Outcome: Number of Participants With Infection
Description: The investigators will continue to monitor the patients for development of an acute postoperative infection. A deep infection refers to an infection below the superficial soft tissue and likely involving the prosthesis. This will be evaluated by the musculoskeletal infection society consensus on total joint infection.
  Criteria include:(Either one major criteria or four minor criteria) Major criteria Sinus track communicating with the prosthesis Two separate cultures from the joint positive for the same organism
  Minor criteria Elevated erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) Elevated synovial leukocyte count Elevated synovial neutrophil percentage Purulent drainage from the joint One positive fluid culture from the joint Histological analysis of tissue showing more than 5 neutrophils per high power field in 5 fields
Time Frame: (Single point evaluation)-6 weeks post surgery visit
Population: Measured all that enrolled and completed the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PREVENA Group | Standard Group
Number analyzed (Participants) | 7 | 9
Participants
  Deep Infection | 0 | 0
  No deep infection | 7 | 9

ADVERSE EVENTS:
Time Frame: Patients that enrolled in the study were followed and seen at 2 weeks postoperatively. The study was terminated prior to patients returning for their 6 week visit so they were not seen by the research staff after 2 weeks. All patients were followed by chart review to confirm adverse events within 6 months of enrolling in the study.
Description: Personal examination at 2 weeks, chart review at 6 months.
Arm/Group | PREVENA Group | Standard Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PREVENA Group (N=7) | Standard Group (N=9)
Wound drainage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Wound drainage for 2 weeks postoperatively requiring antibiotics

LIMITATIONS AND CAVEATS:
Major Limitation-Study could not be completed due to the loss of research personnel early during the trial. We did not have the funding to provide for an additional personnel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT02355691/Prot_SAP_000.pdf